CLINICAL TRIAL: NCT00085813
Title: A Phase II, Open-Label Study of Ispinesib in Subjects With Locally Advanced or Metastatic Platinum-Refractory or Platinum-Relapsed Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Ispinesib In Patients With Advanced Or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP20007
Record Dates: First submitted 2004-06-14; First posted 2004-06-17 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Platinum-Refractory; Platinum-Relapsed; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ispinesib

INTERVENTIONS:
Drug: Ispinesib

SUMMARY:
This study was designed to determine how effective and safe Ispinesib is in treating locally advanced or metastatic Non-small Cell Lung cancer in patients who have received a platinum-based chemotherapy and whose disease continues to progress. Treatment involves a 1-hr treatment given intravenously (IV), repeated once every 21 days. A patient may continue treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times over 24 hr period to measure the amount of drug in your body at specific times after the drug is given. Blood samples will also be taken for routine lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have received only one prior platinum-based chemotherapy regimen.
* Blood tests will be done to check if blood counts are adequate for taking part in the study.

Exclusion Criteria:

* Received more than 1 chemotherapy regimen in the past or have less than adequate liver and kidney function.
* Females who are pregnant.
* Any unstable, pre-existing major medical condition or history of other cancers.
* Have received an investigational drug, chemotherapy, radiation treatment or surgery within 28 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Overall Response Rate of tumor.

SECONDARY OUTCOMES:
Safety and tolerability: adverse events, changes from baseline in vital signs and clinical laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (11):
- United States (7):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
- GSK Investigational Site, Sutton, Surrey, United Kingdom